CLINICAL TRIAL: NCT02709239
Title: Prenatal Docosahexaenoic Acid (DHA) & Neurofunctional Development
Brief Title: Prenatal DHA and Neurofunctional Development
Acronym: PANDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00003792; 1R01HD086001 (NIH)
Record Dates: First submitted 2016-03-04; First posted 2016-03-16 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Use and Dose of Prenatal DHA Supplementation
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- DHA 200mg (Active Comparator): Participants will receive 200mg DHA to take per day. Participants will be asked to take four capsules containing 50mg DHA each.
  Interventions: Dietary Supplement: DHA 200mg
- DHA 800mg (Experimental): Participants will receive 800mg DHA to take per day. Participants will be asked to take four capsules containing 200mg DHA each.
  Interventions: Dietary Supplement: DHA 800mg

INTERVENTIONS:
Dietary Supplement: DHA 200mg — 4 50mg capsules of DHA to be taken by mouth daily
  Other Names: Docosahexaenoic Acid
  Arms: DHA 200mg
Dietary Supplement: DHA 800mg — 4 200mg capsules of DHA to be taken by mouth daily
  Other Names: Docosahexaenoic Acid
  Arms: DHA 800mg

SUMMARY:
The purpose of this study is to learn how much DHA to give to mothers in order to provide enough to the baby. Researchers will also learn if there are differences in development of the baby up to 12 months after birth.

DETAILED DESCRIPTION:
Docosahexaenoic acid (DHA) is an essential nutrient. Our bodies make DHA from the foods we eat. If we eat foods with a lot of DHA, like fatty ocean fish, we have more DHA in our bodies. DHA is found in all cells of the body but is especially high in nerve cells of the brain and eye. Babies get DHA from the mother when they're in the womb. After birth, they can get DHA from breast milk or infant formulas.

This study will enroll pregnant women and follow them and their baby until the baby is 12 months old. Changes in the development of the baby will be tracked. Half of the participants in this study will receive 200mg of DHA to take daily. The other half of participants will receive 800mg of DHA to take daily. Participants, along with the researchers, will not know which dose of DHA they are receiving.

ELIGIBILITY:
Inclusion Criteria:

* Women in their 12th to 20th week of gestation
* Participants agree to consume the study capsules from enrollment to delivery
* Healthy weight, overweight and obese women (determined by body mass index; BMI) are eligible
* Must be available by telephone

Exclusion Criteria:

* Underweight women and women who exceed 250 lbs at enrollment
* Women with serious systemic infection, cancer, major organ disease or systemic lupus erythematosus
* Women with multiple infants or fetal diagnosis of congenital cardiac structural or conduction defects or brain malformations
* Diagnosis of Type I diabetes, and/or hypertension
* Reported drug and/or alcohol abuse
* Unwilling to take capsules, or be contacted by phone
* Do not understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Maternal-Infant DHA Equilibrium | Delivery (birth)
  Maternal blood samples and infant cord blood will be collected at delivery and Red Blood Cell (RBC) DHA concentrations between maternal-infant pairs will be compared. Maternal-Infant DHA Equilibrium occurs if newborn cord blood DHA is less than or equal to the mother's DHA at delivery.

SECONDARY OUTCOMES:
Fetal neurodevelopment as indexed by heart rate variability (HRV) and autonomic brain age scores (fABAS) | 32 weeks gestational age
  Group comparisons will be made between time-domain metrics of fetal HRV (SDNN, RMSSD) and fABAS at two time points.
Fetal neurodevelopment as indexed by heart rate variability (HRV) and autonomic brain age scores (fABAS) | 36 weeks gestational age
  Group comparisons will be made between time-domain metrics of fetal HRV (SDNN, RMSSD) and fABAS at two time points.
Infant Neurodevelopment | 1 month postnatal age
  Brain neurophysiology will be measured at 1 month of age. Assessments of band-limited spectral power during resting-state will be assessed. Event-related potentials (ERP) to auditory stimuli will be recorded. Group comparisons will be made between measures of resting state spectral power and auditory ERP components.
Infant Neurodevelopment | 6 months postnatal age
  Brain neurophysiology will be measured at 6 months of age. Assessments of band-limited spectral power during resting-state will be assessed. Event-related potentials (ERP) to visual stimuli will be recorded. Group comparisons will be made between measures of resting state spectral power and visual ERP components.
Infant Neurodevelopment | 12 months postnatal age
  Brain neurophysiology will be measured at 12 months of age. Assessments of band-limited spectral power during resting-state will be assessed. Event-related potentials (ERP) to visual stimuli will be recorded. Group comparisons will be made between measures of resting state spectral power and visual ERP components.
Infant Behavioral Assessment | 4 months postnatal age
  Heart-rate derived attention metrics and ocular latency (eye movements) will be recorded at 4 months.
Infant Behavioral Assessment | 6 months postnatal age
  Heart-rate derived attention metrics and ocular latency (eye movements) will be recorded at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Gustafson, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gustafson KM, Christifano DN, Hoyer D, Schmidt A, Carlson SE, Colombo J, Mathis NB, Sands SA, Chollet-Hinton L, Brown AR, Mudaranthakam DP, Gajewski BJ. Prenatal docosahexaenoic acid effect on maternal-infant DHA-equilibrium and fetal neurodevelopment: a randomized clinical trial. Pediatr Res. 2022 Jul;92(1):255-264. doi: 10.1038/s41390-021-01742-w. Epub 2021 Sep 22. PMID 34552200
- [Derived] Christifano DN, Chollet-Hinton L, Hoyer D, Schmidt A, Gustafson KM. Intake of eggs, choline, lutein, zeaxanthin, and DHA during pregnancy and their relationship to fetal neurodevelopment. Nutr Neurosci. 2023 Aug;26(8):749-755. doi: 10.1080/1028415X.2022.2088944. Epub 2022 Jun 17. PMID 35715980